CLINICAL TRIAL: NCT03866629
Title: The Effect of Lifitegrast On Refractive Accuracy And Symptoms In Dry Eye Patients Undergoing Cataract Surgery
Status: Completed | Type: Observational
Sponsor: MDbackline, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: IIR-USA-001246
Record Dates: First submitted 2018-12-20; First posted 2019-03-07 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — lifitegrast

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lifitegrast 5%: Patients will receive lifitegrast 0.5% eye drops twice daily 4 weeks prior to cataract surgery.
  Interventions: Drug: Lifitegrast

INTERVENTIONS:
Drug: Lifitegrast — Lifitegrast ophthalmic solution 5%

SUMMARY:
To determine if Xiidra® lifitegrast plays a role in the refractive accuracy when administered to patients preoperatively who are scheduled for cataract surgery and have a tear break up time (TBUT) ≤ 10 seconds and central corneal staining as defined by the Oxford scale

DETAILED DESCRIPTION:
This will be a 4-week multicenter investigator-initiated study, in which a maximum of 200 subjects will be enrolled.

As many as two thirds of patients undergoing cataract surgery have dry eye. Often this latter condition is under treated i.e., any dry eye treatment such as artificial tears, that is being pursued in not adequately controlling the visually significant ocular surface disruption, and patient still have corneal staining or a reduced tear break-up time (TBUT).

The investigators hypothesize that lifitegrast administered at least 4-week prior to pre-operative biometry measurements will improve both the quality of measurements used to choose an intraocular lens implant for surgery and the symptoms of patients with this combination of conditions. This finding would suggest that pre-treatment with lifitegrast can improve both the accuracy of surgery and patient comfort.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with planned cataract surgery
2. Central or inferior corneal fluorescein staining defined by the Oxford Scale
3. Reduced tear break up time (TBUT) ≤ 10 seconds.
4. Able to comprehend and sign a statement of informed consent.
5. Willing and able to complete all required postoperative visits.

Exclusion Criteria:

1. Ocular surgery (e.g., intraocular, oculoplastic, corneal or refractive surgical procedure
2. Clinically significant ocular trauma.
3. Active ocular Herpes simplex or Herpes Zoster infection
4. Ocular inflammation (uveitis, iritis, scleritis, episcleritis, keratitis, conjunctivitis) at the discretion of the investigator.
5. Ocular infection (e.g., viral, bacterial, mycobacterial, protozoan or fungal infection or the cornea, conjunctiva, lacrimal gland, lacrimal sac or eyelids including hordeolum/stye).
6. Active, systemic or local disease condition that causes clinically significant ocular surface irritation such that it could interfere with the questions in the survey and examination findings.
7. Moderate to severe (Grade 2-4) allergic, vernal or giant papillary conjunctivitis.
8. Severe (Grade 3 or 4) inflammation of the eyelid (e.g., blepharochalasis, staphylococcal blepharitis or seborrheic blepharitis)
9. Eyelid abnormalities that significantly affect the lid function (e.g., entropion, ectropion, tumor, edema, blepharospasm, lagophthalmos, severe trichiasis, severe ptosis).
10. Ocular surface abnormality that may compromise the corneal integrity (e.g., prior chemical burn, recurrent corneal erosion, corneal epithelial defect, Grade 3 corneal fluorescein staining, map dot fingerprint dystrophy, or the effect of any other ophthalmic medication that might in the opinion of the investigator compromise the ocular surface integrity).
11. Participation in another ophthalmic clinical trial involving a therapeutic drug or device within 30 days prior to enrollment date.
12. Participation in this trial in the same patient's fellow eye
13. Patients who are pregnant or breastfeeding or who may become pregnant during participation in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This will be a multicenter US investigator initiated clinical trial, in which a maximum of 200 eyes will be treated with lifitegrast ophthalmic solution (5%) prior to planned cataract surgery.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
Increase accuracy of preoperative biometry at predicting postoperative equivalent refractive error | 4 weeks
  Increase accuracy of preoperative biometry at predicting postoperative equivalent refractive error after 4 weeks of lifitegrast ophthalmic solution (5%) BID.

SECONDARY OUTCOMES:
Compare SPEED questionnaire scores before and after 4 weeks of lifitegrast treatment | 4 weeks
  To compare the difference in Standard Patient Evaluation of Eye Dryness Questionnaire (SPEED) scores before and after 4 weeks of therapy with lifitegrast BID among patients with signs of significant dry eye (decreased TBUT or corneal staining) with planned cataract surgery. The SPEED questionnaire gives a score from 0 to 28 that is the result of 8 items that assess frequency and severity of symptoms. Speed Score severity rating: 0-4 Mild, 5-7, Moderate, 8+ Severe.
Determine the percentage of patients with low SPEED scores | 4 weeks
  To determine the percentage of patients with low Standard Patient Evaluation of Eye Dryness Questionnaire (SPEED) scores (≤5 seconds) among patients with signs of significant dry eye (decreased TBUT or corneal staining) with planned cataract surgery. To determine whether this sub-group with asymptomatic dry eye experienced a mean improvement in accuracy of biometry readings after 4 weeks of Lifitegrast symptoms. The SPEED questionnaire gives a score from 0 to 28 that is the result of 8 items that assess frequency and severity of symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard Eye Associates, Laguna Hills, California, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual patient data available.

REFERENCES:
- [Result] Behrens A, Doyle JJ, Stern L, Chuck RS, McDonnell PJ, Azar DT, Dua HS, Hom M, Karpecki PM, Laibson PR, Lemp MA, Meisler DM, Del Castillo JM, O'Brien TP, Pflugfelder SC, Rolando M, Schein OD, Seitz B, Tseng SC, van Setten G, Wilson SE, Yiu SC; Dysfunctional tear syndrome study group. Dysfunctional tear syndrome: a Delphi approach to treatment recommendations. Cornea. 2006 Sep;25(8):900-7. doi: 10.1097/01.ico.0000214802.40313.fa. PMID 17102664
- [Result] Geerling G, Tauber J, Baudouin C, Goto E, Matsumoto Y, O'Brien T, Rolando M, Tsubota K, Nichols KK. The international workshop on meibomian gland dysfunction: report of the subcommittee on management and treatment of meibomian gland dysfunction. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):2050-64. doi: 10.1167/iovs.10-6997g. No abstract available. PMID 21450919